CLINICAL TRIAL: NCT02331485
Title: RANDOMISED CONTROL STUDY TO ASSES THE ROLE OF NEGATIVE PRESSURE WOUND THERAPY (NPWT) IN THE MANAGEMENT OF WOUND IN SURGICAL PATIENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St James Connolly Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sebastian Smolarek, M.D, St James Connolly Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NPWT Ireland
Record Dates: First submitted 2014-08-04; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Wound Infection; Wound Complication
Keywords: Prevention of wound infection and wound complication
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICO + Acticoat group (Experimental): Patients randomized to negative pressure group will received negative pressure dressing (Pico Wound Management System - manufacture by Smith & Nephew) associated with Acticoat Flex dressing which will be applied immediately after skin closure in a conventional way and left in place for 7 days. Negative pressure dressing will be changed once during 7 days period - after day 2 to 4. Wound complications within first 30 days of surgery will be recorded on clinical examination.
  Interventions: Device: PICO + Acticoat group
- Standard Wound management (Active Comparator): If a patient is randomized to standard wound treatment group - he/she will receive standard skin closure and standard Mepore dressing, which will be changed on a daily basis.
  Interventions: Device: PICO + Acticoat group

INTERVENTIONS:
Device: PICO + Acticoat group — Comparison between Pico and Acticoat dressing change after 3 and 7 days with standard Mepor dressing change on daily basis.
  Other Names: PICO; Acticoat Flexi 7 dressing

SUMMARY:
Aim of the study is to assess the role of negative pressure therapy in the prevention of the complication of the laparotomy wound in the high risk patients group.

Primary outcome: Reduction in wound infection rate by 50%

Secondary outcome: Reduction of the length of hospital stay Decrease of using abx. for wound management Decrease cost of patient treatment

DETAILED DESCRIPTION:
Wound complications are common in general surgical patients after laparotomy. The rate of Surgical Site Infections after elective surgery ranges between 3-30%, depending of the study.

There are subgroups of patients with co-morbid conditions that put them at high risk of wound complications. These co-morbid conditions include increase BMI, known malignancy, diabetes mellitus, emergency surgery, malnutrition, smoking and diffuse atherosclerotic disease involving arteries. Management of these complicated wounds are a significant source of psychological trauma to patients and significantly increases hospital stay and cost.

Since its introduction, Negative Pressure Wound Therapy (NPWT) has been used mainly to deal with chronic wounds. Mechanism of action of NPWT includes protection of wound bed, splinting of soft tissues, reduction of oedema, increasing blood perfusion of wound and enhancing granulation tissue. Application of Negative Pressure Wound Therapy to prevent wound complications is a new concept, which has been successfully applied in acute wounds in orthopaedics, gynecological and cardiothoracic surgery patients.

There is limited data about the use of Negative Pressure Wound Therapy in high risk general surgical patients with acute wounds, but available studies suggest significant reduction in wound complication rate and hospital costs. There is a need for a randomised controlled study to assess the reduction of wound complication ratio.

Patient will be randomized to two groups:

Group 1. Standard wound treatment, Group 2. Treatment with negative pressure wound therapy (NPWT). If a patient is randomized to standard wound treatment group - he/she will receive standard skin closure and standard Mepore dressing, which will be changed on a daily basis.

Patients randomized to negative pressure group will received negative pressure dressing (Pico Wound Management System - manufacture by Smith & Nephew) associated with Acticoat Flex dressing which will be applied immediately after skin closure in a conventional way and left in place for 7 days. Negative pressure dressing will be changed once during 7 days period - after day 2 to 4. Wound complications within first 30 days of surgery will be recorded on clinical examination.

Participants will be recruited from patients undergoing elective and emergency surgery in Connolly Hospital, Beaumont Hospital, St Vincent University Hospital and Mater Misericordiae University Hospital based on inclusion or exclusion criteria.

Inclusion criteria:

1. One from below:

   * High BMI
   * Malignancy
   * Malnutrition
   * T2 DM
   * Emergency surgery
   * Post radio chemotherapy
   * On steroids
   * Open colorectal resection
2. At least two from below:

   * Smoking
   * Age>75
   * Diffuse atherosclerotic disease involving arteries

Exclusion criteria:

* Low risk laparotomy wound (none of the above criteria)
* Age < 18

Patient who fulfills inclusion criteria will be contacted prior to surgery by a research team member. Details of the study and risks and benefits will be explained to the patient. After obtaining consent the patient will be randomized to one of two groups - standard wound treatment or negative pressure treatment - by senior research team member. depending on the randomisation patient will recived appropriate dressing. Surgical wound will be asses on day 2 to 4, on day 7 and on day 30. Prior to first dressing application, after 2-4 days and on day 30 a wound swap will be obtain for C&S. Any wound complication will be recorded in research evaluation form.

ELIGIBILITY:
Inclusion Criteria:

1. One from below:

   * High BMI
   * Malignancy
   * Malnutrition
   * T2 DM
   * Emergency surgery
   * Post radio chemotherapy
   * On steroids
   * Open colorectal resection
2. At least two from below:

   * Smoking
   * Age>75
   * Diffuse atherosclerotic disease involving arteries

Exclusion Criteria:

* Low risk laparotomy wound (none of the above criteria)
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Reduction in wound infection by 50% | 1 year

SECONDARY OUTCOMES:
Reduction of the length of hospital stay | 1 year
Decrease antibiotics use in a wound infection management | 1 year
To decrease the cost of patient treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian K Smolarek, M.D, Principal Investigator — Connolly Hospital/Mater Misericordiae University Hospital; Thomas N Walsh, Professor, M.D, FRCSI, Study Chair — Connolly Hospital, Royal College of Surgeons in Ireland
Locations (1):
- Connolly Hospital, Dublin, Ireland

REFERENCES:
- [Background] Lewis LS, Convery PA, Bolac CS, Valea FA, Lowery WJ, Havrilesky LJ. Cost of care using prophylactic negative pressure wound vacuum on closed laparotomy incisions. Gynecol Oncol. 2014 Mar;132(3):684-9. doi: 10.1016/j.ygyno.2014.01.014. Epub 2014 Jan 17. PMID 24440649
- [Background] Ousey KJ, Atkinson RA, Williamson JB, Lui S. Negative pressure wound therapy (NPWT) for spinal wounds: a systematic review. Spine J. 2013 Oct;13(10):1393-405. doi: 10.1016/j.spinee.2013.06.040. Epub 2013 Aug 24. PMID 23981819
- [Background] Hansen E, Durinka JB, Costanzo JA, Austin MS, Deirmengian GK. Negative pressure wound therapy is associated with resolution of incisional drainage in most wounds after hip arthroplasty. Clin Orthop Relat Res. 2013 Oct;471(10):3230-6. doi: 10.1007/s11999-013-2937-3. PMID 23539123
- [Background] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014
- [Background] Stoffan AP, Ricca R, Lien C, Quigley S, Linden BC. Use of negative pressure wound therapy for abdominal wounds in neonates and infants. J Pediatr Surg. 2012 Aug;47(8):1555-9. doi: 10.1016/j.jpedsurg.2012.01.014. PMID 22901916